CLINICAL TRIAL: NCT01278849
Title: A Multi-center, Open-label, Dose-escalation Study to Assess the Pharmacokinetics of ASA404 in Adult Cancer Patients With Impaired Hepatic Function and With Normal Hepatic Function
Brief Title: An Open-label, Dose Escalation Study to Assess the Pharmacokinetics of of ASA404 in Adult Cancer Patients With Impaired Hepatic Function
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CASA404A2105; EudraCT 2009-016471-30 (Registry Identifier: EudraCT)
Record Dates: First submitted 2011-01-17; First posted 2011-01-19 (Estimated); Last update posted 2020-12-09 (Actual); Status verified 2012-11

CONDITIONS: Histologically-proven and Radiologically-confirmed Solid Tumors
Keywords: Advanced or metastatic cancer,; refractory,; core phase,; extension phase,; dose escalation,; standard chemotherapy,; pharmacokinetics,; doctaxel,; paclitaxel,; carboplatin,; safety,; tolerability,; hepatic impairment
MeSH Terms: conditions — Neoplasm Metastasis | interventions — vadimezan

ARMS (1):
- ASA404 + standard therpy (Experimental)
  Interventions: Drug: ASA404

INTERVENTIONS:
Drug: ASA404

SUMMARY:
This study is designed to obtain pharmacokinetic data following a single-dose 20-minute i.v. administration of ASA404 (900, 1200, or 1800 mg/m2) in adult cancer patients with varying degrees of hepatic impairment. The study will be carried out in cancer volunteer patients (utilizing controls with normal hepatic function) who will be assigned to four hepatic impairment groups according to their pre-dose (Day-1) and total bilirubin level. The study will consist of two phases, a (Core Phase) that will evaluate the pharmacokinetics of a single i.v. dose (900, 1200 and 1800 mg/m2) of ASA404 in adult cancer patients with impaired hepatic function, and compared to controls with normal hepatic function. The assessments will be done on the safety and tolerability of that single dose in adult cancer patients with impaired hepatic function and compared to controls with normal hepatic function. The Extension Phase will consist of assessing the safety and tolerability of ASA404 at the same three doses in combination with a sponsor-approved taxane-based regimen in adult cancer patients with impaired hepatic function and compared to controls with normal hepatic function.

ELIGIBILITY:
Inclusion Criteria:

* Patients having histologically-proven solid tumors, who are refractory to standard chemotherapy;
* Patients whom chemotherapy with an investigational agent in combination with docetaxel, or paclitaxel + carboplatin is appropriate;
* Age ≥ 18 years old
* Creatinine clearance according to Cockcroft-Gault formula ≥ 60 mL/min
* A minimum of 4 weeks must have elapsed since the last treatment with other cancer therapies;
* Potassium, calcium, magnesium and phosphorus values within the normal range Total bilirubin ≤ 6 X ULN

Exclusion Criteria:

* Patients having CNS metastases, must have a CT or MRI of the brain performed to rule out CNS metastases;
* Patients with leptomeningeal disease metastases;
* Major surgery </ 4 weeks prior to the start of study;
* Prior exposure to VDAs or other vascular targeting agents;
* Right bundle branch block (RBBB), complete left bundle branch block (LBBB);
* Administration of CYP1A2 and CYP3A4/5 enzyme inducing or inhibiting drugs within 14 days prior to starting study drug;

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2010-01; Primary Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
(Core Phase)To evaluate the PK of a single intravenous dose (900, 1200 and 1800 mg/m2) of ASA404 in adult cancer patients with impaired hepatic function compared to matching patients with normal hepatic function | 18 months

SECONDARY OUTCOMES:
To assess the safety and tolerability of a single i.v. dose (900, 1200 and 1800 mg/m2) of ASA404 in adult cancer patients with impaired hepatic function as compared to controls with normal hepatic function | 18 months
(Extension Phase) assess the safety & tolerability of ASA404 either alone or in combination with a sponsor approved taxane-based regimen in adult cancer patients with impaired hepatic function as compared to controls with normal hepatic function | 18 months
To assess the safety of the combined regimen on the frequency and severity of adverse events and the number of laboratory values worsening from baseline based on the CTCAE grade assessment. | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Investigative Site
Locations (4):
- Italy (2):
  - Novartis Investigative Site, Ancona, AN
  - Novartis Investigative Site, Milan
- New Zealand (2):
  - Novarts Investigative Site, Auckland
  - Novartis Investigative Site, Wellington

REFERENCES:
- See also: Results for CASA404A2105 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=5164